CLINICAL TRIAL: NCT03245502
Title: The Effect of Blood Transfusion on Venoarterial PCO2 Difference in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Turkiye Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Büşra Tezcan, Specialist doctor, Turkiye Yuksek Ihtisas Education and Research Hospital
Other Study IDs: 1297
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Cardiac Procedure Complication
Keywords: tissue oxygenation
MeSH Terms: interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transfused: Patients who have blood transfusion during cardiac surgery
  Interventions: Biological: Blood transfusion
- Not-Transfused: Patients who don't have blood transfusion during cardiac surgery

INTERVENTIONS:
Biological: Blood transfusion — The transfusion of erythrocyte suspension
  Groups: Transfused

SUMMARY:
Venoarterial CO2 difference(delta PCO2), lactate, central venous oxygen saturation(ScVO2) will be recorded in several steps in coronary artery bypass graft and valvular cardiac operations. The patients will be divided into two groups as Transfused, and Non-Transfused Groups observationally. The trend of delta CO2, lactate, ScVO2, postoperative creatinine values, postoperative complications and 28 days mortality will be compared.

DETAILED DESCRIPTION:
Preoperative creatinine values, demographic data, comorbidities will be recorded in ASA I-II elective coronary artery and valvular cardiac surgery patients. Intraoperative delta PCO2, lactate, ScVO2 will be recorded in several steps. The patients will be divided into two groups as Transfused, and Non-Transfused Groups observationally. The trend of delta CO2, lactate, ScVO2, postoperative creatinine values, postoperative complications and 28 days mortality will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery, stable cardiac function

Exclusion Criteria:

* Clinical signs of heart failure, symptomatic cerebral or peripheral failure, uncontrolled diabetes mellitus

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 18-75 years cardiac surgery patients
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Complication | 5 days
  The postoperative neurologic, renal, hepatic, respiratory complications

SECONDARY OUTCOMES:
Mortality | 28 days
  mortality

CONTACTS AND LOCATIONS:
Overall Officials: Demet Bölükbaşı, Specialist, Study Chair — Turkiye Yuksek Ihtisas Education and Research Hospital; Sema Turan, Asc prof, Study Director — Turkiye Yuksek Ihtisas Education and Research Hospital; Dilek Kazancı, Asc prof, Study Chair — Turkiye Yuksek Ihtisas Education and Research Hospital; Sultan Sevim Yakın, Specialist, Study Chair — Turkiye Yuksek Ihtisas Education and Research Hospital; Hija Yazıcıoğlu, Asc Prof, Study Chair — Turkiye Yuksek Ihtisas Education and Research Hospital; Aysegül Özgok, Prof, Study Director — Turkiye Yuksek Ihtisas Education and Research Hospital
Locations (1):
- Turkiye Yuksek Ihtisas Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No